CLINICAL TRIAL: NCT03706313
Title: A Comparison of Analgesic Efficacy of Ultrasound-guided Genicular Nerve Block Versus Saline Injection for Total Knee Replacement: a Prospective, Randomized Controlled Trial
Brief Title: Genicular Nerve Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00100879
Record Dates: First submitted 2018-10-11; First posted 2018-10-15 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Post-operative Pain
Keywords: Total knee replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genicular nerve block with bupivacaine (Active Comparator): The ultrasound-guided genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler will be used to identify the arterial structures which serve as landmarks for the corresponding nerves.
  After skin local anesthetic infiltration, a 10 cm 21G insulated block needle will be inserted and aligned with the ultrasound scanning plane. Once satisfactory position of the needle is confirmed, 5mL of a solution containing 15 ml 0.25% bupivacaine with 2mg dexamethasone or 5mL saline will be slowly injected. Spread of local anesthetic will be documented adjacent to the target nerve. This procedure will be performed at the site of the three genicular nerves described.
  Interventions: Drug: 15mL 0.25% bupivacaine; Procedure: Genicular nerve block
- Genicular nerve block with saline (Placebo Comparator): The ultrasound-guided genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler will be used to identify the arterial structures which serve as landmarks for the corresponding nerves.
  After skin local anesthetic infiltration, a 10 cm 21G insulated block needle will be inserted and aligned with the ultrasound scanning plane (in-plane approach). Once satisfactory position of the needle time is confirmed, 5mL of a saline will be slowly injected. Spread of local anesthetic will be documented adjacent to the target nerve. This procedure will be performed at the site of the three genicular nerves described.
  Interventions: Procedure: Genicular nerve block; Drug: Saline

INTERVENTIONS:
Drug: 15mL 0.25% bupivacaine — Patients will be randomly assigned to either a genicular nerve block with bupivacaine or saline
  Arms: Genicular nerve block with bupivacaine
Procedure: Genicular nerve block — The ultrasound-guided genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. Color Doppler will be used to identify the arterial structures which serve as landmarks for the corresponding nerves.
  After skin local anesthetic infiltration, a 10 cm 21G insulated block needle will be inserted and aligned with the ultrasound scanning plane. Once satisfactory position of the needle is confirmed, 5mL of a solution containing 15 ml of 0.25% bupivacaine with 2mg dexamethasone or 5mL saline will be slowly injected. Spread of local anesthetic will be documented adjacent to the target nerve. This procedure will be performed at the site of the three genicular nerves described.
Drug: Saline — Patients will be randomly assigned to either a genicular nerve block with bupivacaine or saline
  Arms: Genicular nerve block with saline

SUMMARY:
This study seeks to examine the analgesic efficacy of genicular nerve blocks for pain after total knee replacement.

DETAILED DESCRIPTION:
Part of the way in which pain is controlled during total knee replacement surgery is through a nerve block. The investigators have developed an effective protocol for pain control after knee replacement, but know that many patients still experience pain around the knee after knee replacement. There are nerves around the knee that carry pain impulses from behind the knee. The investigators believe that placing numbing medicine around these nerves can help with pain in front of the knee after surgery, in addition to the standard nerve block placed for knee replacement surgery. This may result in taking less pain medication by mouth,and having less pain with movement. For this study, before the operation, either a placebo solution or the local anesthetic bupivacaine (a numbing solution) will be placed at three sites around the knee where these nerves reside. The investigators will evaluate how participants feel in recovery after surgery, during the stay in the hospital, and call at home one week after surgery. Knowing if numbing these nerves helps with pain after surgery will help us further refine our postoperative care plan for patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for primary elective total knee arthroplasty
* American Society of Anesthesiologists Physical Status I-III
* BMI 18-40 kg/m2

Exclusion Criteria:

* Inability to cooperate with protocol
* Inability to understand or speak English
* Allergy to ropivacaine, bupivacaine or other local anesthetic
* Contraindication to peripheral nerve block (e.g. local infection, neurologic deficit or disorder, previous trauma or surgery to ipsilateral knee, etc.)
* Revision knee surgery
* Chronic opioid consumption (daily morphine equivalent of >30 mg for at least four weeks prior to surgery)
* History of chronic pain
* History of psychiatric disorder
* History of diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Gadsden, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rambhia M, Chen A, Kumar AH, Bullock WM, Bolognesi M, Gadsden J. Ultrasound-guided genicular nerve blocks following total knee arthroplasty: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2021 Oct;46(10):862-866. doi: 10.1136/rapm-2021-102667. Epub 2021 Jul 14. PMID 34261807

RESULTS

PARTICIPANT FLOW:
Groups:
- Genicular Nerve Block With Bupivacaine and Dexamethasone: The ultrasound-guided genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. 5 mL of 0.25% bupivacaine 0.67 mg dexamethasone will be administered at each of the 3 genicular nerves.
- Genicular Nerve Block With Saline: The ultrasound-guided sham genicular nerve block will be performed at the site of the superior lateral, the superior medial, and the inferior medial genicular nerves. 5 mL of 0.9% normal saline will be administered at each of the 3 genicular nerves.
Period: Overall Study
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.9 (6.8) | 67.1 (7.6) | 68.9 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 17
  Male | 10 | 13 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Height [Mean (Standard Deviation); unit: cm] | 171.1 (10.0) | 170.4 (11.3) | 170.7 (10.5)
Weight [Mean (Standard Deviation); unit: kg] | 86.5 (19.8) | 87.2 (17.5) | 86.8 (18.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m∧2] | 29.3 (4.7) | 30.0 (5.3) | 29.7 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption at 24 Hours Post-op
Description: Opioid consumption documented in medical recorded will be converted to oral morphine equivalents.
Time Frame: 24 hours after operation
Measure: Mean (Standard Deviation); unit: milligrams of oral morphine equivalents
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
milligrams of oral morphine equivalents | 22.9 (19.8) | 58.1 (34.8)

2. Secondary Outcome: Worst Pain Rating Score (NRS-11) at Rest on Postoperative Day 1
Description: The Numerical Rating Scale (NRS) is an 11-point numeric rating scale, with 0 representing "no pain" and 10 "unbearable pain." This scale demonstrates reliability and validity and is widely used to assess acute pain after surgery.
Time Frame: Postoperative Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 2.7 (1.9) | 3.5 (1.6)

3. Secondary Outcome: Worst Pain Rating Score (NRS-11) With Movement on Postoperative Day 1
Description: as for outcome 2
Time Frame: Postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 4.9 (2.4) | 6.3 (1.9)

4. Secondary Outcome: Total Opioid Consumption Through 48 Hours
Description: Total of all opioids consumed converted to oral morphine equivalents.
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: milligrams of oral morphine equivalents
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
milligrams of oral morphine equivalents | 50.3 (39.8) | 97.6 (56.2)

5. Secondary Outcome: Opioid Consumption on Postoperative Day 7
Description: Self-reported (by telephone questionnaire) opioid consumption in oral morphine equivalents on postoperative day 7
Time Frame: Postoperative day 7
Measure: Mean (Standard Deviation); unit: milligrams of oral morphine equivalents
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
milligrams of oral morphine equivalents | 10.4 (13.7) | 22.6 (24.2)

6. Secondary Outcome: Worst Pain Rating Score (NRS-11) on Postoperative Day 7
Description: as for outcome 2
Time Frame: Postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 4.4 (2.0) | 5.0 (2.2)

7. Secondary Outcome: Sleep Quality Measured by Number of Times Awakened by Pain During the First Postoperative Night
Description: The patient will be questioned by a member of the research team about how many times they were awoken by pain overnight.
Time Frame: Postoperative day 1
Measure: Median (Full Range); unit: number of times awoken by pain
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
number of times awoken by pain | 0 [0 to 3] | 1 [0 to 4]

8. Secondary Outcome: Patient Satisfaction With Pain Control at 24 h
Description: Patient reported satisfaction with his/her pain control at 24 h on a scale of 0-10 (0=completely dissatisfied, 10=completely satisfied)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 9.1 (0.9) | 8.6 (1.1)

9. Secondary Outcome: Patient Satisfaction With Pain Control on Postoperative Day 7
Description: Patient reported satisfaction with his/her pain control on postoperative day 7 on a scale of 0-10 (0=completely dissatisfied, 10=completely satisfied)
Time Frame: Postoperative day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
score on a scale | 8.8 (1.6) | 8.9 (1.2)

10. Secondary Outcome: 20 Meter Walk Test Time Performed on Postoperative Day 1
Description: This standardized test measures the time it takes for the participant to walk 20 meters at their usual walking pace. The 20-meter walk test is a physical function measure commonly used in clinical research studies and rehabilitation clinics to measure gait speed and monitor changes in patients' physical function over time.
Time Frame: On postoperative day 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
Number analyzed (Participants) | 20 | 20
seconds | 74.2 (40.8) | 80.2 (43.6)

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Genicular Nerve Block With Bupivacaine and Dexamethasone | Genicular Nerve Block With Saline
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/13/NCT03706313/Prot_SAP_000.pdf